CLINICAL TRIAL: NCT03532815
Title: A Randomized Controlled Trial of Lifestyle Intervention for Cardiovascular Disease Risk Factors Among Female Residents at the National Guard Residential City, Jeddah, Saudi Arabia, 2015
Brief Title: Lifestyle Intervention for Cardiovascular Disease Risk Factors Among Female Residents at the National Guard Residential City, Jeddah, Saudi Arabia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: King Abdullah International Medical Research Center (Other)
Responsible Party: Principal Investigator, Jumana Khouja, Assistant Consultant, King Abdullah International Medical Research Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: RJ13/039/J
Record Dates: First submitted 2017-12-06; First posted 2018-05-22 (Actual); Last update posted 2019-11-06 (Actual); Status verified 2019-11

CONDITIONS: Cardiovascular Diseases
Keywords: Cardiovascular Diseases, Framingham risk score, Life style modification, Randomized Controlled Trial
MeSH Terms: conditions — Cardiovascular Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Lifestyle Modification group (Active Comparator)
  Interventions: Behavioral: Lifestyle Modification
- Control group (No Intervention)

INTERVENTIONS:
Behavioral: Lifestyle Modification
  Arms: Lifestyle Modification group

SUMMARY:
Cardiovascular disease (CVD) remains the major cause of mortality globally. Applying a comprehensive interventional program based on the individual's risk may reduce the incidence and complications of CVD; thus, helping to decrease the burden on the healthcare system. This study compared the effects of a 3-month intervention involving lifestyle modification and physical activity with standard care in women ≥30 years having a moderate-to-high risk of CVD, with respect to improving physical activity and cardiovascular disease risk factors at the National Guard Residential City in Jeddah, Saudi Arabia, in 2015. The effects of this community-based lifestyle program were assessed through a randomized controlled trial. Women in the intervention group (n=31) received health education, exercise training, and diet counselling as individuals and in groups according to the participant's risk. Women in the control group (n=28) received one health education session at the screening site. The Framingham risk score (FRS) was calculated at baseline and at 3 months for both groups. The mean participant age was 42±8 years.

ELIGIBILITY:
Inclusion Criteria:

1. Women aged ≥ 30 years.
2. The participants must be at moderate to high-risk of CVD according to FRS.

Exclusion Criteria:

1. Women aged < 30 years.
2. Women aged ≥ 30 years with low risk of CVD according to FRS.
3. Pregnant women.
4. Female patients diagnosed with CVD.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 85 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-08-01 (Actual); Study Completion 2015-09-01 (Actual)

PRIMARY OUTCOMES:
Framingham Risk Scores Reduction | 3 months
  The proportion of individuals with moderate Framingham risk scores (FRS) reducing their risk by 10% and the proportion of individuals with high (FRS) reducing their risk by 25% using the Framingham risk score. It consists of six point scores including age, total cholesterol, smoking status, HDL level, diabetes status, systolic Blood Pressure and Treatment Status. The sum of these points will result in an estimate of the 10-Year risk of developing cardiovascular event and for risk categorization of low (< 10% FRS), moderate (10%-19% FRS), or high risk (≥ 20% FRS).

SECONDARY OUTCOMES:
Framingham Risk Category Changes | 3 months
  The proportion of individuals reducing their risk by ≥ 1 risk category using the Framingham risk score. It consists of six point scores including age, total cholesterol, smoking status, HDL level, diabetes status, systolic Blood Pressure and Treatment Status. The sum of these points will result in an estimate of the 10-Year risk of developing cardiovascular event and for risk categorization of low (< 10% FRS), moderate (10%-19% FRS), or high risk (≥ 20% FRS). .

CONTACTS AND LOCATIONS:
Overall Officials: Jumana Khouja, MD, SBCM, Principal Investigator — KAIMRC

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Cox JL, Vallis TM, Pfammatter A, Szpilfogel C, Carr B, O'Neill BJ. A novel approach to cardiovascular health by optimizing risk management (ANCHOR): behavioural modification in primary care effectively reduces global risk. Can J Cardiol. 2013 Nov;29(11):1400-7. doi: 10.1016/j.cjca.2013.03.007. Epub 2013 Jun 21. PMID 23796526
- Available data/document: Study Protocol — https://sites.google.com/view/lifestyle-intervention-/home

DOCUMENTS (1):
  • Study Protocol (2018-07-08): https://cdn.clinicaltrials.gov/large-docs/15/NCT03532815/Prot_001.pdf